CLINICAL TRIAL: NCT01012869
Title: AngiographiC Evaluation of the Everolimus-Eluting Stent in Chronic Total Occlusions - the ACE-CTO Study
Acronym: ACE-CTO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Emmanouil S. Brilakis, MD, PhD, VA North Texas Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-070
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Occlusions
Keywords: Coronary chronic total occlusions
MeSH Terms: conditions — Coronary Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- everolimus-eluting stent (Experimental): patients undergoing treatment of a coronary chronic total occlusion (at least 3-months old) using everolimus-eluting stents (Xience, Abbott Vascular) or Promus (Boston Scientific)
  Interventions: Device: everolimus-eluting stent

INTERVENTIONS:
Device: everolimus-eluting stent — everolimus-eluting stent (Xience, Abbott Vascular) or Promus (Boston Scientific)

SUMMARY:
Chronically total occlusions (CTO) are difficult to treat and have high risk for restenosis. Although everolimus-eluting stents (EES) [(Xience, Abbott Vascular) or Promus (Boston Scientific)] are very promising for the treatment of CTOs due to their low late loss and excellent deliverability, there are currently no published data on EES implantation in CTOs.

The specific aim of this proposal is to examine the 8-month incidence of binary angiographic in-stent restenosis (defined as a stenosis of > 50% of the minimum lumen diameter of the target stent) after implantation of the EES in CTO.

It is the investigators hypothesis that EES-treated CTO lesions will have ≤ 20% 8-month in-stent binary angiographic restenosis rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Successful treatment of a native coronary artery CTO (defined as a lesion with 100% angiographic stenosis that is at least 3 months old as estimated by clinical information, sequential angiographic information, or both) using everolimus-eluting stents
3. Able and willing to return for angiographic follow-up after 8 months and to be followed clinically for 12 months
4. Agree to participate and provide informed consent

Exclusion Criteria:

1. Planned non-cardiac surgery within the following 12 months
2. Recent positive pregnancy test, breast-feeding, or possibility of a future pregnancy
3. Coexisting conditions that limit life expectancy to less than 12 months
4. Patients who have a creatinine above 2.5 mg/dL (unless they require hemodialysis, in which case they are eligible to participate)
5. History of an allergic reaction or significant sensitivity to everolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
In-stent binary angiographic restenosis rate | 8 months

SECONDARY OUTCOMES:
In-stent neointimal hyperplasia, as assessed by intravascular ultrasonography | 8 months
Percent stent strut coverage, as assessed by optical coherence tomography | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Principal Investigator — North Texas Veterans Healthcare System; Subhash Banerjee, MD, Study Director — North Texas Veterans Healthcare System
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Kotsia A, Navara R, Michael TT, Sherbet DP, Roesle M, Christopoulos G, Rangan BV, Haagen D, Garcia S, Maniu C, Pershad A, Abdullah SM, Hastings JL, Kumbhani DJ, Luna M, Addo T, Banerjee S, Brilakis ES. The AngiographiC Evaluation of the Everolimus-Eluting Stent in Chronic Total Occlusion (ACE-CTO) Study. J Invasive Cardiol. 2015 Sep;27(9):393-400. PMID 26332874